CLINICAL TRIAL: NCT00221754
Title: Pravastatin in HIV-Infected Patients Treated With Highly Active Antiretroviral Therapy
Brief Title: Pravastatin and Protease Inhibitors in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9268-02; 2001-026
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: HIV Infection; Hypercholesterolemia
Keywords: HIV,; protease inhibitors; pravastatin; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hypercholesterolemia | interventions — Pravastatin; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pravastatin (drug)

SUMMARY:
To assess the use of pravastatin in hypercholesterolemic HIV-infected patients treated with protease inhibitors in a randomised double blind study.

DETAILED DESCRIPTION:
Background. Highly Active AntiRetroviral Therapy including protease inhibitors is associated with elevated plasma lipid levels.

Design. randomized double-blind, multicentric.

Intervention. Pravastatin versus placebo for 12 weeks.

Eligibility criteria. Positive for anti-VIH antibodies, stable antiretroviral therapy including at least one PI for >= 3 months, plasma HIV-RNA level of < 50 copies/mL for >= 3 months before randomization, total cholesterol >= 5.5 mmol/L with LDL-cholesterol >= 3.4 mmol/L on fasting status after three months of standardized dietary advice, written informed consent

Outcomes. HIV RNA at 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* confirmed HIV-1 infection (ELISA confirmed by Western-Blot test) ;
* Age above 18 years
* Stable antiretroviral therapy including at least one PI for >= 3 months,
* Plasma HIV-RNA level of < 50 copies/mL for >= 3 months before randomization,
* Total cholesterol > = 5.5 mmol/L with LDL-cholesterol > = 3.4 mmol/L on fasting status after three months of standardized dietary advice,
* signed informed consent

Exclusion Criteria:

* Current AIDS event or infectious disease
* Tumoral, inflammatory, muscle diseases; kidney or hepatic failure
* Psychiatric conditions
* Biological elevated muscular enzymes
* Chronic alcohol consumption
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-03; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
HIV RNA | at 12 weeks

SECONDARY OUTCOMES:
Lipid biological markers
Plasma level of protease inhibitors
CD4 count at 12 weeks
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice BONNET, Dr, Principal Investigator — University Hospital Bordeaux, France; Geneviève CHENE, Pr, Study Chair — University Hospital, Bordeaux France
Locations (1):
- Hôpital Saint André, Service de médecine interne et maladies infectieuses, Bordeaux, France